CLINICAL TRIAL: NCT01440686
Title: A Dose Block-randomized, Double-blinded, Placebo-controlled, Single-dose, Dose-escalation Study to Assess the Safety, Pharmacokinetics and Pharmacodynamics of HL-032 in Healthy Male Volunteers
Brief Title: Safety, Pharmacokinetics and Pharmacodynamics Study of HL-032 in Healthy Male Volunteers
Acronym: HL-032
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: HanAll BioPharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HGR10I_1
Record Dates: First submitted 2011-09-23; First posted 2011-09-26 (Estimated); Last update posted 2012-10-16 (Estimated); Status verified 2012-10

CONDITIONS: Growth Hormone Deficiency
Keywords: Pharmacokinetics; Pharmacodynamics; Safety; Male
MeSH Terms: conditions — Dwarfism, Pituitary | interventions — Human Growth Hormone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- HL-032 30mg (Experimental): A single dose 30mg administered orally
  Interventions: Drug: Somatropin; Drug: Placebo
- HL-032 60mg (Experimental): A single dose 60mg administered orally
  Interventions: Drug: Somatropin; Drug: Placebo
- HL-032 120mg (Experimental): A single dose 120mg administered orally
  Interventions: Drug: Somatropin; Drug: Placebo

INTERVENTIONS:
Drug: Somatropin — A single dose 5.0mg administered subcutaneously(under the skin) via Genotropin
Drug: Placebo — Tablets, oral administrations

SUMMARY:
The purpose of this study is to evaluate the safety, pharmacokinetics and pharmacodynamics of HL-032 after oral administration in healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects
* Age(yr)between 19 and 50
* Signed written informed consent

Exclusion Criteria:

* Known hypersensitivity to Octreotide or hGH(human growth hormone)
* History of Cardiovascular, Respiratory, Renal/Genitourinary, Gastrointestinal, Neurological/Psychic, cancer
* Alcoholic, smokers or drug abusers
* Other conditions which in the opinion of the investigator preclude enrollment into the study

Ages: 19 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2011-09; Primary Completion 2011-12 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Area under the serum hGH(human growth hormone)concentration-time curve | From 0 to the time of the last quantifiable concentration over a 32-hour sampling period
Maximum observed serum hGH concentration | Over a 32-hour sampling period

SECONDARY OUTCOMES:
Area under the effect(IGF-1, IGFBP-3, NEFA)curve | From time 0 to the time of the last concentration(AUECO-t) over 32-hour sampling period
Maximum IGF-1, IGFBP-3, NEFA effect | Over a 32-hour sampling period

CONTACTS AND LOCATIONS:
Overall Officials: Kyung-Sang Yu, Medicine, Principal Investigator — Seoul National University Hospital,Clinical Trial Center/ Clinical Research Institute
Locations (1):
- Seoul National University Hospital,Clinical Trial Center/ Clinical Research Institute, Seoul, South Korea